CLINICAL TRIAL: NCT03760887
Title: A Follow-up Comparison of Sensory Discrimination in Patients With Low Back Pain: a Randomized Control Trial
Brief Title: A Follow-up Comparison of Sensory Discrimination in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Kevin Farrell, Professor, Chair of Clinical Residency Program in Orthopaedic Physical Therapy, St. Ambrose University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StAmbroseU sensory
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2018-11

CONDITIONS: Low Back Pain
Keywords: Low back pain; Sensory; Tactile; Education
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: Patients were randomly assigned to one of two groups (control or experimental).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Home Sensory training (Sham Comparator): Patients who perform a home exercise program only
  Interventions: Other: Home exercise program only
- Home sensory training (Experimental): Patients who perform home exercise and home sensory training
  Interventions: Other: Home exercise program and home program of sensory discrimination

INTERVENTIONS:
Other: Home exercise program only — After 5 minutes of sensory discrimination (using a 9 point grid) in the clinic patients will perform a home exercise program only
  Arms: No Home Sensory training
Other: Home exercise program and home program of sensory discrimination — After 5 minutes of sensory discrimination (using a 9 point grid) in the clinic patients will perform a home exercise program and two 5 minutes sessions of sensory training at home each day.
  Arms: Home sensory training

SUMMARY:
To determine if there is any carry over difference with sensation training to the low back for patients with low back pain with the addition of a training at home. This will be looked at to see if there is a difference in pain or back / leg movement right after the training and in a few days after doing some exercises at home.

DETAILED DESCRIPTION:
In a previous case series patients with chronic Low Back Pain (LBP) who received tactile acuity training to their lower back in the absence of movement, experienced immediate positive changes in pain ratings and spinal movements. These changes, however, where only measured immediate post-intervention. This study aims to use a similar design of sensory discrimination for LBP, but will include a sensory discrimination home exercise program and compare groups at a follow-up visit for any difference between groups (48-96 hours) of the immediate changes. Changes will be assessed for pain and back and leg movement.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 18
* patients presenting at PT with a primary complaint of LBP
* LBP being present for 3 months or more
* fluent in English
* willing to participate in the study
* They also will need someone who can assist with a sensory discrimination HEP.

Exclusion Criteria:

* under age 18
* not able to read/understand the English language
* prisoners
* no medical issues precluding physical therapy treatment (red flags)
* if they had undergone spinal surgery
* if they had any skin or medical condition preventing them from receiving tactile stimuli on the lower back or had specific movement-based precautions, i.e., no active spinal flexion. - Patients presenting with leg pain only
* Patients with neurological deficit only in the lower extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Low Back Pain Rating | Change from baseline to following treatment immediately upon completion of initial session
  Numeric Pain Rating Scale for Back pain (0 = no pain and 10 = worst pain)
Low Back Pain Rating | Change from end of treatment initial session to 2-4 days
  Numeric Pain Rating Scale for Back pain (0 = no pain and 10 = worst pain)
Lumbar Flexion | Change from baseline to treatment immediately upon completion of initial session
  Active trunk forward flexion measured in cm (finger tips to floor)
Lumbar Flexion | Change from end of treatment initial session to 2-4 days
  Active trunk forward flexion measured in cm (finger tips to floor)
Straight Leg Raise | Change from baseline to treatment immediately upon completion of initial session
  Neurodynamic measurement of leg raise (lower limb tension test)
Straight Leg Raise | Change from end of treatment initial session to 2-4 days
  Neurodynamic measurement of leg raise (lower limb tension test)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Farrell, Principal Investigator — St. Ambrose University
Locations (1):
- St. Ambrose university, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louw A, Farrell K, Wettach L, Uhl J, Majkowski K, Welding M (2015) Immediate effects of sensory discrimination for chronic low back pain: a case series. New Zealand Journal of Physiotherapy 43(2)